CLINICAL TRIAL: NCT03770260
Title: MLN9708 (Ixazomib) and MLN4924 (Pevonedistat) in Relapsed/Refractory Multiple Myeloma Patients: A Phase 1b Trial
Brief Title: Ixazomib and Pevonedistat in Treating Patients With Multiple Myeloma That Has Come Back or Does Not Respond to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-03121; NCI-2018-03121 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10249 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10249 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib citrate, pevonedistat) (Experimental): Patients receive ixazomib citrate PO QD on days 1, 8, and 15 of each cycle and pevonedistat IV over 60 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib Citrate; Drug: Pevonedistat

INTERVENTIONS:
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924

SUMMARY:
This phase Ib trial studies side effects and best dose of pevonedistat when given together with ixazomib in treating patients with multiple myeloma that has come back or does not respond to treatment. Pevonedistat and ixazomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of MLN4924 (pevonedistat) in combination with MLN9708 (ixazomib citrate [ixazomib]) in relapsed and/or refractory multiple myeloma (RRMM) patients after more than one previous line of treatment. (Dose-escalation phase) II. Describe the safety profile and tolerability of the combination of MLN9708 (ixazomib) and MLN4924 (pevonedistat) in the proteasome inhibitor (PI)-sensitive and PI-refractory populations. (Dose-expansion phase) III. Determine the anti-tumor activity and overall response rates (ORR) in patients with RRMM with the use of MLN9708 (ixazomib) and MLN4924 (pevonedistat) in combination. (Dose-expansion phase)

SECONDARY OBJECTIVE:

I. Attain pharmacokinetic (PK) characterization of MLN4924 (pevonedistat) in combination with MLN9708 (ixazomib) for the purpose of understanding concentration-effect relationships of both agents. (Dose-escalation phase)

EXPLORATORY OBJECTIVE:

I. To correlate and predict disease response using the following tests: NAD(P)H dehydrogenase (quinone) 1 (NQO1) and cystine/glutamate transporter (SLC7A11) (nuclear factor [erythroid-derived 2]-like 2 [NRF2] target genes): evaluated on whole blood as markers of MLN4924 (pevonedistat) activity.

OUTLINE: This is a dose-escalation study of pevonedistat.

Patients receive ixazomib citrate orally (PO) once daily (QD) on days 1, 8, and 15 of each cycle and pevonedistat intravenously (IV) over 60 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 2-3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have RRMM with measurable disease, as defined by at least one of the following:

  * Serum monoclonal protein >= 0.5 g/dL
  * Urinary monoclonal protein excretion of >= 200 mg/24 hours
  * Kappa or lambda light chain level >= 10 mg/dL with an abnormal free light chain ratio
* At least two prior lines of therapy and all patients should have at least been exposed to a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and an anti-CD38 antibody.

  * For proteasome-sensitive expansion cohort: Patients with MM who relapsed or are refractory to a prior line of therapy not including a proteasome inhibitor
  * For proteasome-relapsed/refractory expansion cohort: Patients with MM who have relapsed after prior PI exposure or are PI-refractory, defined as nonresponsive to treatment or progresses within 60 days of last exposure to a PI
* Age >= 18 years

  * Because no dosing or adverse event (AE) data are currently available on the use of MLN4924 (pevonedistat) in combination with MLN9708 (ixazomib) in patients < 18 years of age, and as this disease is exceptionally uncommon in this age group, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Bilirubin =< institutional upper limit of normal (ULN).

  * Patients with Gilbert's syndrome may enroll if direct bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN
* Creatinine clearance (CrCl) by Cockcroft-Gault >= 30 mL/min
* Known human immunodeficiency virus (HIV) positive patients who meet the following criteria will be considered eligible:

  * CD 4 count > 350 cells/mm^3
  * Undetectable viral load
  * Maintained on modern therapeutic regimens utilizing non-CYP-interactive agents (e.g. excluding ritonavir)
  * No history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections
* The effects of MLN4924 (pevonedistat) and MLN9708 (ixazomib) on the developing human fetus are unknown. For this reason and because NAE inhibitory agents are known to be teratogenic, women of child-bearing potential and men must meet the following criteria:

  * Female patients who are:

    * Postmenopausal for at least one year before the screening visit, OR
    * Surgically sterile, OR
    * If of childbearing potential, agree to practice 1 highly effective method and 1 additional (barrier) method of contraception, at the same time, from the time of signing the informed consent until 4 months after the last dose of the ixazomib and pevonedistat (female and male condoms should not be used together), or agree to abstain from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject (Periodic abstinence [e.g,, calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception)
  * Male patients, even if surgically sterilized, who:

    * Agree to practice effective barrier contraception during the entire time enrolled on study through 4 months after completion of ixazomib and pevonedistat administration (female and male condoms should not be used together), OR
    * Agree to abstain from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception)
  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection
* Patients who are receiving any other investigational agents, within 30 days of the start of this trial and throughout the duration of this trial
* Patients with known central nervous system involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other AEs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN4924 (pevonedistat) or MLN9708 (ixazomib) (including boron or boron-containing products)
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because MLN4924 (pevonedistat) is an NAE inhibitory agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with MLN4924 (pevonedistat), breastfeeding should be discontinued if the mother is treated with MLN4924 (pevonedistat). These potential risks may also apply to the use of MLN9708 (ixazomib) in this study
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period
* Patients with uncontrolled coagulopathy or bleeding disorder
* Known hepatic impairment as defined by known hepatic cirrhosis, hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection

  * Note: Patients who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load
* Known cardiopulmonary disease defined as:

  * Unstable angina;
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV);
  * Myocardial infarction within 6 months prior to first dose (patients who had ischemic heart disease such as acute coronary syndrome [ACS], myocardial infarction, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll);
  * Symptomatic cardiomyopathy
  * Clinically significant arrhythmia:

    * History of polymorphic ventricular fibrillation or torsade de pointes,
    * Permanent atrial fibrillation, defined as continuous atrial fibrillation for >= 6 months,
    * Persistent atrial fibrillation, defined as sustained atrial fibrillation lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening,
    * Grade 3 atrial fibrillation defined as symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation in the past 6 months and
    * Patients with paroxysmal atrial fibrillation or grade < 3 atrial fibrillation for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen
  * Clinically significant pulmonary hypertension requiring pharmacologic therapy
* Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mmHg, diastolic blood pressure > 95 mmHg)
* Prolonged rate corrected QT (QTc) interval >= 500 msec, calculated according to institutional guidelines
* Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram
* Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 (ixazomib), including difficulty swallowing
* Peripheral neuropathy that is grade >= 3, or grade 2 with pain on clinical examination during the screening period
* Patients that have previously been treated with MLN9708 (ixazomib)
* Systemic treatment, within 14 days before the first dose of MLN9708 (ixazomib), with strong CYP3A inducers (rifampin, rifapentine, rifabutin, ritonavir, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort. Clinically significant metabolic enzyme inducers are not permitted during this study
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708 (ixazomib)
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s)
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Joseph, Principal Investigator — Emory University
Locations (9):
- United States (9):
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Pevonedistat 20 mg/meter squared given by infusion and ixazomib 4 mg taken by mouth on days 1, 8 and 15 of every 28-day cycle.
- Dose Level 2: Pevonedistat 40 mg/meter squared given by infusion and ixazomib 4 mg taken by mouth on days 1, 8 and 15 of every 28-day cycle.
- Dose Level 3: Pevonedistat 60 mg/meter squared given by infusion and ixazomib 4 mg taken by mouth on days 1, 8 and 15 of every 28-day cycle.
- Dose Expansion: Pevonedistat at the maximum tolerated dose determined in the dose levels given by infusion and ixazomib 4 mg taken by mouth on days 1, 8 and 15 of every 28-day cycle.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Expansion
Started | 3 | 4 | 1 | 0
Completed | 3 | 3 | 1 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: Pevonedistat 20 mg/m^2 given by a vein in the arm and ixazomib 4 mg taken by mouth on days 1, 8 and 15 of every 28-day cycle.
- Dose Level 2: Pevonedistat 40 mg/m^2 given by a vein in the arm and ixazomib 4 mg taken by mouth on days 1, 8 and 15 of every 28-day cycle.
- Dose Level 3: Pevonedistat 60 mg/m^2 given by a vein in the arm and ixazomib 4 mg taken by mouth on days 1, 8 and 15 of every 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 3 | 4 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 0 | 4
  >=65 years | 0 | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 1 | 3
  White | 0 | 1 | 0 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity (Dose Escalation)
Description: Number of participants experiencing a dose limiting toxicity to determine the maximum tolerated dose (MTD)
Time Frame: At Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1; Dose Level 3: Patients receive pevonedistat 20 mg/meter squared by infusion and ixazomib citrate 4 mg by mouth on days 1, 8, and 15 of each 28-day cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Dose Level 2: Patients receive pevonedistat 40 mg/meter squared by infusion and ixazomib citrate 4 mg by mouth on days 1, 8, and 15 of each 28-day cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 3 | 4 | 1
Participants
  Experienced a Dose Limiting Toxicity | 0 | 0 | 0
  Did Not Experience a Dose Limiting Toxicity | 3 | 3 | 1
  Withdrew from Treatment | 0 | 1 | 0

2. Primary Outcome: Number of Participants Experiencing a Grade 3-5 Adverse Event (Dose Expansion)
Description: Number of participants who experienced a grade 3-5 adverse event in the dose expansion group
Time Frame: Up to 2 years after Treatment
Population: Did not complete dose escalation phase to enroll to the dose expansion phase.
Groups:
- Dose Expansion: Patients receive pevonedistat the maximum tolerated dose (MTD) as determined in the dose escalation phase by infusion ande ixazomib citrate 4 mg by mouth on days 1, 8, and 15 of each 28-day cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

3. Primary Outcome: Overall Response Rate (Dose Expansion)
Description: To determine the overall responses in patients receiving pevonedistat and ixazomib
Time Frame: Up to 2 Years after Treatment
Population: The dose escalation phase was not completed in order to enroll to the dose expansion phase
Arm/Group | Dose Expansion
Number analyzed (Participants) | 0

4. Secondary Outcome: Characterize the Pharmacokinetics (PK) of Pevonedistat and Ixazomib (Dose Escalation)
Description: To understand the concentration-effect relationship of both agents when taken together
Time Frame: Up to 3 months
Population: This data was not collected.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years and 2 months
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/4 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=4) | Dose Level 3 (N=1)
Non-cardiac Chest Pain (General disorders) | 1 | 0 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=4) | Dose Level 3 (N=1)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1
BUN elevated (Blood and lymphatic system disorders) | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1
Fever (General disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 4 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 2 | 1
Weight loss (Investigations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
carpel tunnel repair (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lower Leg Cramping (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Alteration in Breathing Pattern (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blisters (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Enrollment was stopped by the drug company during the third dose level of the Dose Escalation Phase. They discontinued clinical trials using pevonedistat. No participants were enrolled to the Dose Expansion Phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03770260/Prot_SAP_000.pdf
  • Informed Consent Form: P10249_A08ConsentEscalation(Redacted) (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03770260/ICF_001.pdf
  • Informed Consent Form: P10249_A08ConsentExpansion(Redacted) (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03770260/ICF_002.pdf